CLINICAL TRIAL: NCT05006690
Title: Comparison of the Effects of Telerehabilitation and Face-to-Face Clinical Pilates-Based Exercise Training in Individuals With Axial Spondyloarthritis
Brief Title: Telerehabilitation and Face-to-Face Clinical Pilates-Based Exercise in Individuals With Axial Spondyloarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Nur Banu Karaca, Research Assistant, Physiotherapist, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA-21035
Record Dates: First submitted 2021-08-08; First posted 2021-08-16 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Axial Spondyloarthritis; Ankylosing Spondylitis
Keywords: spinal stabilization exercise; telerehabilitation; clinical pilates; Ankylosing spondylitis; Axial spondyloarthritis; biopsychosocial
MeSH Terms: conditions — Axial Spondyloarthritis; Spondylitis, Ankylosing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telerehabilitation Training Group (Experimental): In the telerehabilitation group, an individualized rehabilitation program according to the principles of clinical pilates exercises based on spinal stabilization will be applied via video conference, 3 days a week, 1 hour, online in real-time, accompanied by a physiotherapist, for 8 weeks.
  In the first session, informative training about the disease (pathophysiology of axial spondyloarthritis, its course, physical structures it covers, etc.), pain management training (information about the relationship between pain, muscle spasm, stress, depression, methods that can be used for coping with pain, etc.), exercise. The importance of exercise training (trunk stabilization, anatomy) and aims will be given within the scope of patient education.
  Interventions: Other: Clinical Pilates-Based Exercise Training
- Face-to-Face Training Group (Experimental): In the face-to-face training group, an individualized rehabilitation program according to the principles of clinical pilates exercises based on spinal stabilization will be applied in the clinic under the supervision of a physiotherapist for 1 hour, 3 days a week, for 8 weeks.
  In the first session, informative training about the disease (pathophysiology of axial spondyloarthritis, its course, physical structures it covers, etc.), pain management training (information about the relationship between pain, muscle spasm, stress, depression, methods that can be used for coping with pain, etc.), exercise. The importance of exercise training (trunk stabilization, anatomy) and aims will be given within the scope of patient education.
  Interventions: Other: Clinical Pilates-Based Exercise Training

INTERVENTIONS:
Other: Clinical Pilates-Based Exercise Training — Clinical Pilates-Based exercise training based on spinal stabilization aim at controlling the position of the trunk over the pelvis to provide optimal energy production and energy transfer to distal segments and involve the cocontraction of muscles, which may restore stability to the spine.

SUMMARY:
Spondyloarthritis (SpA) refers to a group of rheumatic diseases that share common clinical, genetic and imaging features. They are divided into two: axial (axSpA) and peripheral. In addition to the pain caused by sacroiliitis and spondylitis, which are the main complaints, patients often experience joint stiffness, fatigue, mood disturbances and various degrees of functional limitations, and the quality of life of individuals can be significantly affected. Although there is consensus about the positive effects of exercise in AxSpA, no exercise regimen has been shown to be superior to another. Another exercise model whose effectiveness has been researched in recent years is "clinical pilates exercises". It is a version of the Pilates exercises created by Joseph Pilates, modified by physiotherapists to emphasize the most valuable components in the diagnosis and management of injuries and to increase their safety. Clinical Pilates exercises are an exercise model based on spinal stabilization principles. In addition, it has the principles of awareness, balance, breathing, concentration, centering, control, efficiency, flow, sensitivity, isolation and harmony. There are many studies investigating the effects of these exercises in the field of rehabilitation and highlighting improvements in different diseases, including ankylosing spondylitis, which is considered the prototype of axSpA. No study has been found examining exercise training applied via telerehabilitation to individuals with AxSpA and its effects. The aim of this study is to compare the effects of telerehabilitation and face-to-face clinical pilates-based exercise training on individuals with axial spondyloarthritis. Volunteers who meet the inclusion criteria will be randomly divided into 'telerehabilitation training group' and 'face-to-face training group' using the sealed envelope method. The individualized rehabilitation program will be applied to each group for 1 hour, 3 days a week, for 8 weeks. Disease-specific performance measurements and patient-reported scales that evaluate patients' disease activity, functionality, mood, quality of life, fear-avoidance, levels and perceptions of the disease will be applied to individuals three times in total: at the beginning, after the 8-week rehabilitation program and 6 months after the second evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with axial spondyloarthritis
* Between the ages of 18-65,
* Literate,
* Having sufficient smartphone/computer knowledge to participate in the study or having a relative who can help in this regard,
* Having a smart phone/computer and an active internet connection,
* Individuals who have not exercised regularly in at least the last 3 months will be included in the study.

Exclusion Criteria:

* Having a diagnosis of uncontrolled/clinically significant other disease (chronic obstructive pulmonary disease, congestive heart failure, endocrine system diseases, neurological, psychological diseases, etc.),
* Malignancies
* Having a history of previous surgery on the spine and extremities and therefore loss of function,
* Pregnant individuals,
* Continuing another rehabilitation program,
* Have other conditions that prevent exercise,
* A significant change in medication regimen occurs while the study is ongoing,
* Individuals who do not agree to participate in the study and do not give written consent will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-12-18 (Actual); Primary Completion 2025-08-19 (Actual); Study Completion 2025-08-19 (Actual)

PRIMARY OUTCOMES:
Evaluation of Functional Level | 5 minutes, through study completion, an average of 8 weeks, change from baseline functional level at 8 weeks.
  Bath Ankylosing Spondylitis Functional Index (BASFI): The index consists of 10 questions in total. For each item, the patient marks the VAS consisting of a 100 mm line. The score range is 0-100. The Turkish version study was conducted by Karatepe et al. made by. A high score indicates a bad result.
Evaluation of Disease Activity | 3 minutes, through study completion, an average of 8 weeks, change from baseline disease activity at 8 weeks.
  Bath Ankylosing Spondylitis Disease Activity Index (BASDAI): The index consists of 6 items questioning 5 symptoms in total. The response of each item is evaluated with the Visual Analog Scale (VAS). A total score of ≥ 4 indicates active disease. Turkish version study Akkoç et al. made by.

SECONDARY OUTCOMES:
Evaluation of Spinal Mobility and Hip Function | 10 minutes, through study completion, an average of 8 weeks, change from baseline spinal mobility and hip function at 8 weeks.
  Bath Ankylosing Spondylitis Metrology Index (BASMI): The index, which consists of five clinical measurements, namely cervical rotation, tragus-wall distance, lumbar lateral flexion, modified Schober's test, and intermalleolar distance, is accepted as the most valid method for evaluating the axial skeleton. The higher the BASMI score the more severe the patient's limitation of movement.
Evaluation of Quality of Life | 1 minutes, through study completion, an average of 8 weeks, change from baseline quality of life at 8 weeks.
  Ankylosing spondylitis quality of life questionnaire (ASQoL): ASQoL, which is one of the most commonly used disease-specific scales to measure the quality of life in axspa, consists of 18 items and total score ranges from 0-18. A high score indicates bad quality of life. The Turkish version study was conducted by Duruoz et al. made by.
Evaluation of Biopsychosocial Status | 10 minutes, through study completion, an average of 8 weeks, change from baseline biopsychosocial status at 8 weeks.
  BETY-Biopsychosocial Questionnaire (BETY-BQ): Each of the questions in this scale, which consists of 30 different cognitive belief statements, is scored between 0-4. The total score ranges from 0 to 120. A high score indicates a poor biopsychosocial level. It is a scale developed by Ünal et al.
Evaluation of Depression and Anxiety Levels | 7 minutes, through study completion, an average of 8 weeks, change from baseline depression and anxiety levels at 8 weeks.
  Hospital Anxiety and Depression Scale (HADS):This scale consisting of 14 questions, odd-numbered questions question anxiety and even questions question depression. The options take values between 0-3, with a high score indicating a bad emotional state. The cut-off values of the scale were determined as 10 for the anxiety subscale and 7 for the depression subscale. The Turkish version study was done by Aydemir et al.
Evaluation of Kinesiophobia | 5 minutes, through study completion, an average of 8 weeks, change from baseline kinesiophobia at 8 weeks
  Tampa Kinesophobia Scale (TCS): It is a 17-question scale that evaluates injury avoidance and fear of movement, and Kori et al. developed by. The Turkish version is from Tunca-Yılmaz et al. Made by. Its scoring is scored with "1 = Strongly disagree, 4 = Strongly agree". The score is calculated by reversing items 4, 8, 12, and 16. The total score is between 17 and 68. It is understood that the higher the score, the higher the kinesophobia. A total score of more than 37 is considered to be a high degree of kinesophobia.
Evaluation of Illness Perception | 3 minutes, through study completion, an average of 8 weeks, change from baseline illness perception at 8 weeks.
  Brief Illness Perception Scale (BIPQ): In this scale, which consists of 9 questions, each question evaluates a component of the perception of illness. The first eight questions take values between 0-10. A high score indicates an increased level of perception of the disease as worrisome. The total score ranges from 0 to 80. The ninth question is an open-ended question that questions the patient's opinion about the possible causes of the disease. Turkish validity and reliability study was done by Karataş et al.
Evaluation of Physical Performance | 10-15 minutes, through study completion, an average of 8 weeks, change from baseline physical performance at 8 weeks.
  Ankylosing Spondylitis Performance Index (ASPI): Objective measurement of functional level ASPI consists of standardized performance tests of 3 items evaluated with patient feedback in the BASFI form: (1) picking up 6 pencils one by one by bending forward at the waist; (2) put on socks (3 repetitions); and (3) standing from supine position (3 repetitions). During tests, patients are allowed to use a chair or desk/table to sit or lean on. The time to complete a task is measured and recorded in seconds for each test. Additionally, for each test, test-related pain and effort are recorded with patient-reported scores (numerical rating scale (NRS) and Borg scale, respectively).
Evaluation of rib cage mobility: Chest Expansion Measurement | 2 minutes, through study completion, an average of 8 weeks, change from baseline chest expansion at 8 weeks.
  Chest expansion is an ASAS recommended assessment to measure rib cage mobility. The patient is asked to place his hands behind his head. Chest circumference is measured at the fourth intercostal space during maximal inspiration and maximal expiration. Two repetitions are made and the better value is recorded.
Side Bridge Endurance Test: Evaluation of spinal stabilization | Testing time depends on the patient, through study completion, an average of 8 weeks, change from baseline spinal stabilization at 8 weeks.
  Side bridge tests are measured by recording the time in seconds in which the patient maintains the position in which he/she is lying on his/her side on the mat, extending both legs straight and lifting his hips off the mat with the support he receives from his elbows and feet. The test is terminated when the person cannot maintain this position. Both sides are measured and averaged.
Exercise Self-Efficacy Scale (ESES): Assessment of exercise self-efficacy | 5 minutes, through study completion, an average of 8 weeks, change from baseline self-efficacy at 8 weeks.
  The ESES scale, developed by Bandura (1997), consists of 18 items that question a person's beliefs about their competence in exercising. The participant scores his/her self-confidence between 0 and 100 for each item asked. The validity and reliability of the scale in Turkish was conducted by Bozkurt et al.
ASAS (Assessment of SpondyloArthritis International Society) Health Index (ASAS-HI): Evaluation of health and disability | 5 minutes, through study completion, an average of 8 weeks, change from baseline disability at 8 weeks.
  The ASAS Health Index was developed by the International Society for the Assessment of SpondyloArthritis (ASAS) to assess the health of patients with all forms of spondyloarthritis (especially radiographic and non-radiographic axial SpA). It is a self-report survey and measures functionality and health in patients with 17 questions. It has Turkish validity and reliability.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Faculty of Physical Therapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No